CLINICAL TRIAL: NCT02021396
Title: Benefit of Prophylactic Embolization of the Splenic Salvage in Trauma Patients at High Risk of Splenectomy.
Brief Title: Benefit of Prophylactic Embolization of the Splenic Salvage
Acronym: Splash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DCIC 13 02
Record Dates: First submitted 2013-12-03; First posted 2013-12-27 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Splenic Trauma
Keywords: splenic rescue; splenectomy
MeSH Terms: interventions — Embolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Embolization (Experimental): this arm of the study was interventional (embolization) with CT scans at inclusion (D0, to validate the inclusion criteria), at one month (D30-validating the primary endpoint) and at 6 months (D180) read by 2 expert radiologists blinded to the study arm
  Interventions: Procedure: Embolization
- Surveillance (No Intervention): this arm of the study was non-interventional (surveillance), with CT scans at inclusion (D0, to validate the inclusion criteria), at one month (D30-validating the primary endpoint) and at 6 months (D180 ) read by 2 expert radiologists blinded to the study arm

INTERVENTIONS:
Procedure: Embolization — this arm of the study was interventional (splenic artery embolization)
  Arms: Embolization

SUMMARY:
The main objective is to show that splenic embolization improves salvage rate at one month in a population of hemostatically stable closed splenic trauma patients with a high risk of splenectomy

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 and under 75 years
* hemodynamically stable patients (systolic BP ≥ 90 mm Hg and no hemorrhagic shock)
* Suffered a closed splenic trauma within the last 48 hours
* A high risk of splenectomy:

  * Reaching spleen Moore grade 4 and 5 in the abdominal injected CT or
  * Reaching spleen Moore 3 and at least one of the following characteristics:

    * Important Hemoperitoneum (when visible in the pelvic area).
    * Severe associated impairment (NISS-New Injury Severity Score greater than or equal to 15)
* Patients volunteering to participate in the study, having signed the consent form or with the agreement of the family if the patient is not capable of giving consent; after adequate information and delivery of the patient and/or family information leaflet.
* covered by a social security scheme or beneficiary of such a plan.

Exclusion Criteria:

* Patients whose usual residence is outside the European Economic Community
* Patient with hemodynamic instability (systolic blood pressure <9 despite resuscitation maneuver)
* Patient with open splenic trauma
* Patient with surgical indication excluding the possibility of monitoring splenic trauma
* Patient with an indication for embolization of a body other than the spleen at the time of inclusion
* Patient with an indication for splenic embolization as a result of a post-traumatic vascular anomaly (active leakage of contrast agent, pseudoaneurysm or early splenic arteriovenous fistula).
* Patients aged less than 18 years and ≥ 75 years
* Patients with a previous spleen disease (tumor, infection, vascular anomaly intrasplenically)
* Patient with trauma Moore grade 1 or 2
* Patient with trauma grade Moore 5 with total ischemia of the spleen
* Patients who underwent partial or total splenectomy before inclusion
* Patient having acquired or innate immune deficiency
* All indications not permitting the achievement of embolization
* Pregnant woman
* Person deprived of liberty by judicial or administrative decision, person subject to a measure of legal protection.
* Patient currently participating in a clinical study or having participated in a clinical study in the month preceding the inclusion
* Patient with a condition or a history of mental or psychiatric disorder or any other factor limiting their ability to participate in an informed manner and to comply with the protocol.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-02; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Rescue rate | Splenic Rescue at 30 days
  The main objective is to show that splenic embolization improves salvage rate at one month in a population of hemostatically stable closed splenic trauma patients with a high risk of a splenectomy. The primary endpoint is an immunocompetent spleen i.e. intact or treated by surgical methods for splenic preservation of at least 50% of splenic vascularized tissue in the event of secondary laparotomy or with necrosis of less than 50% by volume. This criterion will be validated by a review of the initial scans by a panel of two senior radiologists blinded to the study arm.

SECONDARY OUTCOMES:
Mortality | At 1 and 6 months
Morbidity | at 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pr Catherine ARVIEUX, Principal Investigator — University Clinic of Digestive Surgery and Emergency
Locations (1):
- University Hospital Grenoble Alpes, Grenoble, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnoletti JP, Karam J, Brodsky J. Early postoperative complications of splenectomy for hematologic disease. Am J Clin Oncol. 1999 Apr;22(2):114-8. doi: 10.1097/00000421-199904000-00002. PMID 10199442
- [Background] Requarth JA, D'Agostino RB Jr, Miller PR. Nonoperative management of adult blunt splenic injury with and without splenic artery embolotherapy: a meta-analysis. J Trauma. 2011 Oct;71(4):898-903; discussion 903. doi: 10.1097/TA.0b013e318227ea50. PMID 21986737
- [Background] Benoist S. [Median and long-term complications of splenectomy]. Ann Chir. 2000 May;125(4):317-24. doi: 10.1016/s0003-3944(00)00201-7. French. PMID 10900732
- [Background] Altamura M, Caradonna L, Amati L, Pellegrino NM, Urgesi G, Miniello S. Splenectomy and sepsis: the role of the spleen in the immune-mediated bacterial clearance. Immunopharmacol Immunotoxicol. 2001 May;23(2):153-61. doi: 10.1081/iph-100103856. PMID 11417844
- [Background] Kotsanas D, Al-Souffi MH, Waxman BP, King RW, Polkinghorne KR, Woolley IJ. Adherence to guidelines for prevention of postsplenectomy sepsis. Age and sex are risk factors: a five-year retrospective review. ANZ J Surg. 2006 Jul;76(7):542-7. doi: 10.1111/j.1445-2197.2006.03775.x. PMID 16813615
- [Background] Bain IM, Kirby RM. 10 year experience of splenic injury: an increasing place for conservative management after blunt trauma. Injury. 1998 Apr;29(3):177-82. doi: 10.1016/s0020-1383(97)00170-8. PMID 9709417
- [Background] Peitzman AB, Heil B, Rivera L, Federle MB, Harbrecht BG, Clancy KD, Croce M, Enderson BL, Morris JA, Shatz D, Meredith JW, Ochoa JB, Fakhry SM, Cushman JG, Minei JP, McCarthy M, Luchette FA, Townsend R, Tinkoff G, Block EF, Ross S, Frykberg ER, Bell RM, Davis F 3rd, Weireter L, Shapiro MB. Blunt splenic injury in adults: Multi-institutional Study of the Eastern Association for the Surgery of Trauma. J Trauma. 2000 Aug;49(2):177-87; discussion 187-9. doi: 10.1097/00005373-200008000-00002. PMID 10963527
- [Background] Haan JM, Biffl W, Knudson MM, Davis KA, Oka T, Majercik S, Dicker R, Marder S, Scalea TM; Western Trauma Association Multi-Institutional Trials Committee. Splenic embolization revisited: a multicenter review. J Trauma. 2004 Mar;56(3):542-7. doi: 10.1097/01.ta.0000114069.73054.45. PMID 15128125
- [Background] Liu PP, Lee WC, Cheng YF, Hsieh PM, Hsieh YM, Tan BL, Chen FC, Huang TC, Tung CC. Use of splenic artery embolization as an adjunct to nonsurgical management of blunt splenic injury. J Trauma. 2004 Apr;56(4):768-72; discussion 773. doi: 10.1097/01.ta.0000129646.14777.ff. PMID 15187739
- [Background] Gaarder C, Dormagen JB, Eken T, Skaga NO, Klow NE, Pillgram-Larsen J, Buanes T, Naess PA. Nonoperative management of splenic injuries: improved results with angioembolization. J Trauma. 2006 Jul;61(1):192-8. doi: 10.1097/01.ta.0000223466.62589.d9. PMID 16832270
- [Background] Sabe AA, Claridge JA, Rosenblum DI, Lie K, Malangoni MA. The effects of splenic artery embolization on nonoperative management of blunt splenic injury: a 16-year experience. J Trauma. 2009 Sep;67(3):565-72; discussion 571-2. doi: 10.1097/TA.0b013e3181b17010. PMID 19741401
- [Background] Ekeh AP, McCarthy MC, Woods RJ, Haley E. Complications arising from splenic embolization after blunt splenic trauma. Am J Surg. 2005 Mar;189(3):335-9. doi: 10.1016/j.amjsurg.2004.11.033. PMID 15792763
- [Background] Haan J, Bochicchio G, Kramer M, Scalea T. Air following splenic embolization: infection or incidental finding? Am Surg. 2003 Dec;69(12):1036-9; discussion 1039-40. PMID 14700287
- [Background] Bessoud B, Duchosal MA, Siegrist CA, Schlegel S, Doenz F, Calmes JM, Qanadli SD, Schnyder P, Denys A. Proximal splenic artery embolization for blunt splenic injury: clinical, immunologic, and ultrasound-Doppler follow-up. J Trauma. 2007 Jun;62(6):1481-6. doi: 10.1097/TA.0b013e318047dfb8. PMID 17563670
- [Background] Sugg SL, Gerndt SJ, Hamilton BJ, Francis IR, Taheri PA, Rodriguez JL. Pseudoaneurysms of the intraparenchymal splenic artery after blunt abdominal trauma: a complication of nonoperative therapy and its management. J Trauma. 1995 Sep;39(3):593-5. doi: 10.1097/00005373-199509000-00034. PMID 7473932
- [Background] Jacquot S, Boyer O. [Heterogeneity and function of human B lymphocytes]. Med Sci (Paris). 2006 Dec;22(12):1075-80. doi: 10.1051/medsci/200622121075. French. PMID 17156729
- [Background] Ozturk H, Dokucu AI, Onen A, Otcu S, Gedik S, Azal OF. Non-operative management of isolated solid organ injuries due to blunt abdominal trauma in children: a fifteen-year experience. Eur J Pediatr Surg. 2004 Feb;14(1):29-34. doi: 10.1055/s-2004-815777. PMID 15024676
- [Background] Stevenson M, Segui-Gomez M, Lescohier I, Di Scala C, McDonald-Smith G. An overview of the injury severity score and the new injury severity score. Inj Prev. 2001 Mar;7(1):10-3. doi: 10.1136/ip.7.1.10. PMID 11289527
- [Background] Moore EE, Cogbill TH, Jurkovich GJ, Shackford SR, Malangoni MA, Champion HR. Organ injury scaling: spleen and liver (1994 revision). J Trauma. 1995 Mar;38(3):323-4. doi: 10.1097/00005373-199503000-00001. No abstract available. PMID 7897707
- [Background] Harbrecht BG, Zenati MS, Ochoa JB, Townsend RN, Puyana JC, Wilson MA, Peitzman AB. Management of adult blunt splenic injuries: comparison between level I and level II trauma centers. J Am Coll Surg. 2004 Feb;198(2):232-9. doi: 10.1016/j.jamcollsurg.2003.10.007. PMID 14759780
- [Background] Burch JM, Ortiz VB, Richardson RJ, Martin RR, Mattox KL, Jordan GL Jr. Abbreviated laparotomy and planned reoperation for critically injured patients. Ann Surg. 1992 May;215(5):476-83; discussion 483-4. doi: 10.1097/00000658-199205000-00010. PMID 1616384
- [Background] Arvieux C. [Visceral traumatology: a necessity in France]. J Chir (Paris). 2003 Oct;140(5):259-60. No abstract available. French. PMID 14631289
- [Background] Brugere C, Arvieux C, Dubuisson V, Guillon F, Sengel C, Bricault I, Regimbeau JM, Pilleul F, Menegaux F, Letoublon C. [Early embolization in the non-operative management of blunt splenic injuries: a retrospective multicenter study]. J Chir (Paris). 2008 Mar-Apr;145(2):126-32. doi: 10.1016/s0021-7697(08)73721-9. French. PMID 18645552
- [Background] Barquist ES, Pizano LR, Feuer W, Pappas PA, McKenney KA, LeBlang SD, Henry RP, Rivas LA, Cohn SM. Inter- and intrarater reliability in computed axial tomographic grading of splenic injury: why so many grading scales? J Trauma. 2004 Feb;56(2):334-8. doi: 10.1097/01.TA.0000052364.71392.70. PMID 14960976
- [Background] Haan JM, Bochicchio GV, Kramer N, Scalea TM. Nonoperative management of blunt splenic injury: a 5-year experience. J Trauma. 2005 Mar;58(3):492-8. doi: 10.1097/01.ta.0000154575.49388.74. PMID 15761342
- [Background] Godley CD, Warren RL, Sheridan RL, McCabe CJ. Nonoperative management of blunt splenic injury in adults: age over 55 years as a powerful indicator for failure. J Am Coll Surg. 1996 Aug;183(2):133-9. PMID 8696544
- [Background] Harbrecht BG. Is anything new in adult blunt splenic trauma? Am J Surg. 2005 Aug;190(2):273-8. doi: 10.1016/j.amjsurg.2005.05.026. PMID 16023445
- [Background] Malangoni MA, Levine AW, Droege EA, Aprahamian C, Condon RE. Management of injury to the spleen in adults. Results of early operation and observation. Ann Surg. 1984 Dec;200(6):702-5. doi: 10.1097/00000658-198412000-00005. PMID 6508398
- [Background] Fingerhut A, Oberlin P, Cotte JL, Aziz L, Etienne JC, Vinson-Bonnet B, Aubert JD, Rea S. Splenic salvage using an absorbable mesh: feasibility, reliability and safety. Br J Surg. 1992 Apr;79(4):325-7. doi: 10.1002/bjs.1800790414. PMID 1576499
- [Background] Madoff DC, Denys A, Wallace MJ, Murthy R, Gupta S, Pillsbury EP, Ahrar K, Bessoud B, Hicks ME. Splenic arterial interventions: anatomy, indications, technical considerations, and potential complications. Radiographics. 2005 Oct;25 Suppl 1:S191-211. doi: 10.1148/rg.25si055504. PMID 16227491
- [Background] Caceres M, Buechter KJ, Tillou A, Shih JA, Liu D, Steeb G. Thoracic packing for uncontrolled bleeding in penetrating thoracic injuries. South Med J. 2004 Jul;97(7):637-41. doi: 10.1097/00007611-200407000-00005. PMID 15301119
- [Background] Steinsapir ES, Coley BD, Fellmeth BD, Roberts AC, Hye RJ. Selective management of iatrogenic femoral artery injuries. J Surg Res. 1993 Jul;55(1):109-13. doi: 10.1006/jsre.1993.1116. PMID 8412076
- [Background] Hagiwara A, Fukushima H, Murata A, Matsuda H, Shimazaki S. Blunt splenic injury: usefulness of transcatheter arterial embolization in patients with a transient response to fluid resuscitation. Radiology. 2005 Apr;235(1):57-64. doi: 10.1148/radiol.2351031132. Epub 2005 Mar 4. PMID 15749973
- [Background] Hiraide A, Yamamoto H, Yahata K, Yoshioka T, Sugimoto T. Delayed rupture of the spleen caused by an intrasplenic pseudoaneurysm following blunt trauma: case report. J Trauma. 1994 May;36(5):743-4. doi: 10.1097/00005373-199405000-00026. PMID 8189480
- [Background] Dror S, Dani BZ, Ur M, Yoram K. Spontaneous thrombosis of a splenic pseudoaneurysm after blunt abdominal trauma. J Trauma. 2002 Aug;53(2):383-5. doi: 10.1097/00005373-200208000-00035. No abstract available. PMID 12169954
- [Background] Owens CA, Alkadri A, Yaghmai B, Warner D, Vitello J. Massive intraperitoneal hemorrhage from traumatic intrasplenic pseudoaneurysms: treatment using superselective embolotherapy. Int Surg. 2001 Oct-Dec;86(4):201-5. PMID 12056461
- [Background] Paya K, Wurm J, Graf M, Pichler P, Oertl M, Mayerhoffer W, Engels M. Intrasplenic posttraumatic pseudoaneurysm secondary to spleen-salvaging surgery. J Trauma. 2002 Apr;52(4):783-5; discussion 785. doi: 10.1097/00005373-200204000-00033. No abstract available. PMID 11956404
- [Background] Oguz B, Cil B, Ekinci S, Karnak I, Akata D, Haliloglu M. Posttraumatic splenic pseudoaneurysm and arteriovenous fistula: diagnosis by computed tomography angiography and treatment by transcatheter embolization. J Pediatr Surg. 2005 Dec;40(12):e43-6. doi: 10.1016/j.jpedsurg.2005.08.003. PMID 16338294
- [Background] Schwartz PE, Sterioff S, Mucha P, Melton LJ 3rd, Offord KP. Postsplenectomy sepsis and mortality in adults. JAMA. 1982 Nov 12;248(18):2279-83. PMID 7131680
- [Background] Waghorn DJ, Mayon-White RT. A study of 42 episodes of overwhelming post-splenectomy infection: is current guidance for asplenic individuals being followed? J Infect. 1997 Nov;35(3):289-94. doi: 10.1016/s0163-4453(97)93232-1. PMID 9459404
- [Background] Holdsworth RJ, Irving AD, Cuschieri A. Postsplenectomy sepsis and its mortality rate: actual versus perceived risks. Br J Surg. 1991 Sep;78(9):1031-8. doi: 10.1002/bjs.1800780904. PMID 1933181
- [Background] Read RC, Finch RG. Prophylaxis after splenectomy. J Antimicrob Chemother. 1994 Jan;33(1):4-6. doi: 10.1093/jac/33.1.4. No abstract available. PMID 8157572
- [Background] Cullingford GL, Watkins DN, Watts AD, Mallon DF. Severe late postsplenectomy infection. Br J Surg. 1991 Jun;78(6):716-21. doi: 10.1002/bjs.1800780626. PMID 2070242
- [Background] Waghorn DJ. Overwhelming infection in asplenic patients: current best practice preventive measures are not being followed. J Clin Pathol. 2001 Mar;54(3):214-8. doi: 10.1136/jcp.54.3.214. PMID 11253134
- [Background] Shih HC, Wang CY, Wen YS, Wu JK, Huang MS, Huang CI, Lee CH. Spleen artery embolization aggravates endotoxin hyporesponse of peripheral blood mononuclear cells in patients with spleen injury. J Trauma. 2010 Mar;68(3):532-7. doi: 10.1097/TA.0b013e3181a7bfaa. PMID 19935106
- [Background] Tominaga GT, Simon FJ Jr, Dandan IS, Schaffer KB, Kraus JF, Kan M, Carlson SR, Moreland S 3rd, Nelson T, Schultz P, Eastman AB. Immunologic function after splenic embolization, is there a difference? J Trauma. 2009 Aug;67(2):289-95. doi: 10.1097/TA.0b013e3181a5e7e2. PMID 19667881
- [Derived] Tidadini F, Martinet E, Quesada JL, Foote A, El Wafir C, Girard E, Arvieux C; SPLASH study group. Patient factors associated with embolization or splenectomy within 30 days of initiating surveillance for splenic trauma. Emerg Radiol. 2024 Dec;31(6):823-833. doi: 10.1007/s10140-024-02285-3. Epub 2024 Oct 4. PMID 39365384
- [Derived] Arvieux C, Frandon J, Tidadini F, Monnin-Bares V, Foote A, Dubuisson V, Lermite E, David JS, Douane F, Tresallet C, Lemoine MC, Rodiere M, Bouzat P, Bosson JL, Vilotitch A, Barbois S, Thony F; Splenic Arterial Embolization to Avoid Splenectomy (SPLASH) Study Group. Effect of Prophylactic Embolization on Patients With Blunt Trauma at High Risk of Splenectomy: A Randomized Clinical Trial. JAMA Surg. 2020 Dec 1;155(12):1102-1111. doi: 10.1001/jamasurg.2020.3672. PMID 32936242